CLINICAL TRIAL: NCT05572398
Title: Translating an In-Person Brief, Bystander Bullying Intervention (STAC) to a Technology-Based - Phase II
Brief Title: Online Bullying Bystander Intervention for Middle Schools Phase II
Acronym: STACII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Boise State University (Other); University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0337; 5R42MD014943 (NIH)
Record Dates: First submitted 2022-09-20; First posted 2022-10-07 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Adolescent; Bullying; Technology; Mental Health
MeSH Terms: conditions — Bullying; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STAC-T (Experimental): STAC-T is a brief technology-based bullying bystander intervention using four strategies: "Stealing the show," "Turning it over," "Accompanying others," and "Coaching compassion." The online curriculum is delivered to middle-school students.
  Interventions: Behavioral: STAC-T
- Assessment Only Control (No Intervention): Assessment Only Control

INTERVENTIONS:
Behavioral: STAC-T — Middle school participants will complete online modules to learn about anti-bullying techniques and bystander intervention.
  Arms: STAC-T

SUMMARY:
School interventions to reduce bullying can be effective but also require substantial time and resources. Online technologies have the potential to deliver effective bullying interventions to a large number of middle school students for less cost. The feasibility of delivering the effective STAC bullying intervention through a mobile web app will be tested using focus groups with middle school students and development and usability testing and the efficacy of the program will be tested using a randomized controlled trial.

DETAILED DESCRIPTION:
While studies support the efficacy of comprehensive, school-wide interventions in reducing bullying, these types of programs can require significant time and financial resources for implementation, resulting in barriers to providing school-based bullying prevention, especially in low-income and rural communities. Additionally, although training bystanders to act as "defenders" on behalf of targets of bullying is an important intervention component, few programs include this as part of their comprehensive strategy. Brief programs that focus on bystander training and require fewer resources are needed to reduce bullying and its negative consequences. The PI (Dr. Midgett) developed STAC, a brief, stand-alone bullying bystander intervention for middle school students, to reduce bullying and mental health risks for bystanders. Brief, in-person programs, however, still pose implementation barrier such as training school personnel, providing external support, and not allowing for large groups of students to be trained at the same time. For this project, the investigators propose to develop a technology-based STAC intervention (STAC-T) that will allow students to customize their experience by selecting avatars and bullying scenarios based on our previous studies conducted in a range of middle schools, including those in low-income and rural communities. The investigators will also incorporate an assessment and personalized feedback component to promote behavior change. The innovative, user-centered design proposed will be inherently sensitive to cultural needs of students and identify personally-appropriate strategies. The specific aims of this application include building the program leveraging our prior work and expertise of an external advisory board, usability and effectiveness testing with middle school students and stakeholders to evaluate feasibility, and testing the efficacy of the program with a randomized controlled trial. The technology-based platform will increase the overall reach, impact, and sustainability of the STAC intervention for bullying prevention. It will substantially reduce cost to increase reach and its interactivity and algorithms can tailor program content to adapt it further for students attending low-income and rural schools. Thus, this low-cost, easy to disseminate technology-based bullying bystander intervention has the potential to have a substantial impact on the problem of bullying and the negative associated consequences for both students who are targets and bystanders in middle school when the problem of bullying peaks. There is a large market for the STAC-T intervention with approximately 100,000 public and private schools with middle-school grades in the United States. Globally, the online education market is growing at 10% a year and the digital health market exceeds $220 billion annually.

ELIGIBILITY:
Inclusion Criteria for Students:

* being enrolled in grades 6, 7, or 8 in a middle/junior high school in Idaho, Oregon, Mississippi, or New Hampshire.
* being selected by school counselors and teachers for having a desire to make a positive difference at school, be mature, and have the ability to positively engage with peers and adults (Aims 1 and 2).
* speaks and reads English or Spanish.
* parent consents and student assents for participation.

Exclusion Criteria for Students:

* participated in a previous study on STAC.
* speaks and reads only a language other than English or Spanish.
* does not consent and/or assent for participation.

Inclusion Criteria for School Personnel:

* employed in a middle/junior high school in Idaho or Mississippi with grades 6, 7, or 8.
* employed as a principal, teacher, or school counselor.
* speaks and reads English or Spanish.
* consents to participate.

Exclusion Criteria for School Personnel:

* participated in a previous study on STAC.
* speaks and reads only a language other than English or Spanish.
* does not consent for participation.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Student-Advocates Pre- and Post-Scale (SAPPS) at Immediate Post-Intervention | Baseline assessment, immediate post-assessment
  An 11-item questionnaire measuring students' knowledge of bullying, knowledge of the STAC-T strategies, and students' confidence to intervene in bullying situations. The minimum value is 0 and the maximum value is 32, and a higher score means a better outcome.
Change from Baseline Student-Advocates Pre- and Post-Scale (SAPPS) at 6 weeks | Baseline assessment, 6-week assessment
  An 11-item questionnaire measuring students' knowledge of bullying, knowledge of the STAC-T strategies, and students' confidence to intervene in bullying situations. The minimum value is 0 and the maximum value is 32, and a higher score means a better outcome.
System Usability Scale (SUS) | Intermediate post-assessment for the randomized trial
  The System Usability Scale is a validated tool for assessing the usability and acceptability of technological products. It is a 10-item questionnaire with 5 response options. The minimum value is 0 and a maximum value is 40. A higher score indicates a perceived ease-of-use from the user.
Change from Baseline Use of Strategies at 6 weeks | Baseline assessment, 6-week assessment
  Questions rating the student's use of each STAC-T strategy using a single item rated on a 5-point Likert scale: "How often would you say you have used these strategies to stop bullying in the past month?" (a) Stealing the Show; (b) Turning it Over; (c) Accompanying Others; and (d) Coaching Compassion.
Change from Baseline Bullying and Cyberbullying Scale for Adolescents (BCS-A) at 6 weeks | Baseline assessment, 6-week assessment
  This questionnaire measures bullying and cyberbullying perpetration and victimization in the past 30 days. The 8-item Bullying Scale assesses bullying perpetration and bullying victimization, and has two sub-scales. The minimum value is 0 and the maximum value is 32, and a higher score means a worse outcome. The 5-item Cyberbullying Scale assesses cyberbullying perpetration and cyberbullying victimization, and has two sub-scales. The minimum value is 0 and the maximum value is 20, and a higher score means a worse outcome.

SECONDARY OUTCOMES:
Center for Epidemiological Studies Depression Scale for Children | Baseline assessment, 6-week assessment
  The 20-item CES-DC measures depressive symptoms in children on a four-point Likert Scale. The minimum value is 0 and the maximum value is 60, and a higher score means a worse outcome.
The Social Avoidance and Distress Scale - General and Fear of Negative Evaluation Scale in the condition Social Anxiety Scale for Adolescents (SAS-A) | Baseline assessment, 6-week assessment
  The 18-item Social Avoidance and Distress Scale - General and Fear of Negative Evaluation Scale will measure anxiety. The minimum value is 0 and the maximum value is 72, and a higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Buller, MA, Principal Investigator — Klein Buendel, Inc.
Locations (2):
- United States (2):
  - Boise State University, Boise, Idaho
  - University of Mississippi, University, Mississippi